CLINICAL TRIAL: NCT04889508
Title: Investigating the Differential Effects of Online Mental Training Interventions on Mental Well-being and Social Cohesion
Brief Title: Investigating Differential Effects of Online Mental Training Interventions on Mental Well-being and Social Cohesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Social Neuroscience Lab (Other)
Collaborators: Charite University, Berlin, Germany (Other); Humboldt-Universität zu Berlin (Other); Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CovSocialPhase2
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Depressive Symptoms; Stress; Empathy; Compassion; Prosocial Behavior; Anxious Symptoms; Loneliness; Resilience; Genetic Markers
MeSH Terms: conditions — Depression; Altruism

STUDY DESIGN:
Masking Description: No masking will be used since both participants and staff need to be aware which condition the participant belongs to in order to be able to attain and provide the appropriate training and practice prior to starting the actual interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Socio-emotional mental training (Experimental): The socio-emotional intervention will consist of 10 weeks of daily Affect Dyad practice with a partner.
  Interventions: Behavioral: Socio-emotional mental training
- Mindfulness-based mental training (Experimental): The intervention will consist of 10 weeks of daily individual Breathing Meditation practice.
  Interventions: Behavioral: Mindfulness-based mental training
- Retest Control Group (Waitlist control) (Other): The retest control group, which is also a waitlist control group, will first not undergo an intervention, but will be tested prior to and after the 10-week period at Pre- and Post-test wherein other groups undergo the interventions.
  In a second step, the waitlist control group will then also undergo a 10-week period of socio-emotional intervention.
  During the first 10-week intervention period, this group will only be tested serving as a re-test control group. After Post-test, however, they will be given the chance to also enroll in a 10-week socio-emotional mental training with the exact same protocol as the socio-emotional intervention experimental group above.
  Both the experimental intervention arm groups will be given the possibility to continue their daily assigned practices (respective socio-emotional and mindfulness-based training exercises) after post-test for the duration of the 10-weeks during which the waitlist control group undergoes the socio-emotional intervention.
  Interventions: Behavioral: Socio-emotional mental training

INTERVENTIONS:
Behavioral: Socio-emotional mental training — Core practice: Affect Dyad. In the Affect Dyad (AD), participants perform a 12-minute partner-based exercise which involves contemplating over one difficult situation and one situation which incurred gratitude in the past 24 hours. Both partners take turns speaking about the two situations while the other partner listens in a non-judgmental manner. While the participants elaborate on the situations, they are asked to focus on the bodily experience of the emotions generated during the situation. The goal of the exercise is to enhance coping with difficult emotions, empathic listening, social sharing, acceptance, and gratitude.
  Arms: Retest Control Group (Waitlist control); Socio-emotional mental training
Behavioral: Mindfulness-based mental training — Core practice: Breathing Meditation. In this intervention, participants will practice 12-minute basic attention-based mindfulness meditation such as the Breathing Meditation (BM). BM is a 12-minute individual exercise that requires participants to focus their attention on the sensations of breathing. Participants have to sustain their attention to breath for long stretches of time, and have to return their attention to their breath when their mind wanders. The key focus is on training attention and interoceptive body awareness. Other practices participants will be taught is mindfulness on sounds (here the object of attention is not the breath but sounds in the environment).
  Arms: Mindfulness-based mental training

SUMMARY:
The SARS-CoV-2 pandemic, and the associated government-imposed isolationary lockdowns, has led to a mental health crisis on a global scale. Empirical studies have reported a drastic increase in mental health problems, such as depression and anxiety, increased loneliness and feelings of disconnectedness from others, while resilience levels have been negatively affected, indicating an urgent need for intervention. The current study study is embedded in a larger study, the CovSocial study (www.covsocial) which focused in its first phase on evaluating the longitudinal changes in vulnerability, resilience and social cohesion during the SARS-CoV-2 pandemic. The present second phase of this CovSocial study will seek to investigate the efficacy of brief online mindfulness-based and socio-emotional interventions in reducing mental health problems, and enhancing psychological resilience, social competencies and social cohesion.

After providing informed consent, participants will be assigned to one of three groups: 1) socio-emotional training group (with Affect Dyads as core exercise), 2) mindfulness-based mental training group (with attention-based mindfulness practices such as Breathing Meditation as core practice), or 3) Retest Control Group (waitlist control).All groups will first undergo a pre-intervention testing phase (pre-test) wherein they will provide a comprehensive baseline measurement which covers psychometric measures (such as questionnaires and behavioral tasks), and biological parameters (saliva samples). During the 10-week intervention period, participants will undergo weekly assessments and daily Ecological Momentary Assessment pre and post the daily exercise practice, using self-report scales and questionnaires delivered through a webapp or mobile app. At the end of the intervention, participants will again undergo an assessment of psychometric measures and biological parameters, same as at pre-intervention time (post-test). In a second portion, the waitlist control group will undergo the socio-emotional intervention and will be tested at post-test II again.

Results will reveal the effectiveness of brief online interventions in enhancing mental health and social cohesion outcomes. In addition to examining pre-post intervention-related changes, we will also use the data from the phase 1 of the project to evaluate the impact of trait markers of and the longitudinal changes in vulnerability, resilience and social cohesion on the intervention-related changes in markers of vulnerability, resilience and social cohesion. We will also evaluate the predictive impact of genetic markers of vulnerability, resilience and social cohesion (assessed in phase 1) on intervention-related changes in our variables of interest.

The present study will serve as a pilot for future application of scalable, low-cost interventions at a broader level to reduce stress, improve mental health and build resilience in the face of global stressors.

ELIGIBILITY:
Inclusion Criteria:

Participants will have to meet the following inclusion criteria:

1. between 18 and 65 years age
2. resident of Berlin
3. proficiency in German.

Exclusion Criteria:

Participants would be excluded:

1. if they do not have access to internet or technical equipment necessary
2. if they have an educational background in psychology
3. if they have regular spiritual practice (including yoga practice with meditative component)
4. if they take medication that influences physiological markers
5. if they have participated in stress reduction programs previously
6. if they suffer from a chronic illness or pain, or if they have a history of or current psychiatric diagnosis.
7. Toronto Alexithymia Scale-20 (TAS-20; exclude if score greater than 60)
8. Patient Health Questionnaire-9 (PHQ-9; exclude if scores greater than 19)
9. Generalized Anxiety Disorder-7 (GAD-7; exclude if scores greater than 15)

Moreover, participants endorsing suicidality on the PHQ-9 will be excluded. Lastly, participants will be further screened for personality disorder on the Standardized Assessment of Severity of Personality Disorder questionnaire and for endorsement of clinical levels of psychological disorder on CID-S.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Beck Depression Inventory (BDI)-II scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring depression symptoms. Higher scores indicate more depression symptoms.
Change from baseline State Trait Anxiety Inventory (STAI) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring state and trait anxiety symptoms. Higher scores indicate more anxiety symptoms.
Change from baseline Connor Davidson Resilience Scale (CDRISC) score at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring psychological resilience. Higher scores indicate more resilience.
Change from baseline UCLA Loneliness Scale at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring loneliness. Higher scores indicate more subjective loneliness.
Change from baseline State Self Compassion Scale (S-SCS) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring compassion towards self. Higher scores indicate more self-compassion.
Change from baseline Perceived Stress Scale (PSS)-10 scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring perceived stress. Higher scores indicate more perceived stress.
Change from baseline Interpersonal Reactivity Index (IRI) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring four aspects of empathy. Higher scores indicate more empathy.
Change from baseline Cortisol Awakening Response at 10 weeks | Assessed at pre-intervention over a period 2 days (Baseline), and then after 10-week intervention period at post-intervention timepoint again for 4 days
  Cortisol Awakening response.
Change from baseline Subjective Stress levels at 10 weeks | Assessed at pre-intervention over a period 8 days (Baseline), and then after 10-week intervention period at post-intervention timepoint again for 8 days
  Assessment of quality of sleep, stressor appraisal, coping with stressor, affective state, valence and temporal orientation of thoughts, perceived emotional control, and interoceptive awareness. Using Ecological Momentary Assessment(EMA).
Change from baseline Brief Resilience Scale (BRS) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring adaptive resilience. Higher scores indicate more resilience.
Change from baseline Difficulties in Emotion Regulation Scale (DERS)-18 scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring difficulties in use of emotion regulation strategies. Higher scores indicate more difficulties in emotion regulation.
Change from baseline Cognitive Emotion Regulation Questionnaire (CERQ)-18 scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring use of emotion regulation strategies. Higher scores on a strategy sub scale indicate more use of the emotion regulation strategy.
Change from baseline Fear of Compassion Scale (FoC) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring fear of compassion towards self. Higher scores indicate more fear of compassion.
Change from baseline Social Value Orientations (SVO) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A task measuring social value orientations and prosocial behavior. Number of choices will be used as the dependent variable.
Change from baseline Zurich Prosocial Game scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A behavioral task assessing levels of prosocial behavior towards others. Number of keys invested in will serve as the dependent variable.
Change from baseline EmpaToM scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A behavioral task assessing empathy and theory of mind. Valence and compassion ratings will serve as the dependent variables.
Change from baseline Social Discounting Task scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A behavioral task assessing prosocial behavior and altruism. The degree of discounting will serve as the dependent variable.
Change from baseline Multidimensional Assessment of Interoceptive Awareness (MAIA) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring interoception. Higher scores indicate more interoceptive awareness.
Change from baseline Sussex-Oxford Compassion Scale (SOC) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring compassion. Higher scores indicate more compassion.
Change from baseline Toronto Alexithymia Scale scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A scale measuring Alexithymia. Higher scores indicate more alexithymia.
Change from baseline Trier Social Stress Test (TSST) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A task assessing cortisol response to social stress. Subjective stress and cortisol levels will serve as the dependent variables.

SECONDARY OUTCOMES:
Change in baseline Dot Probe Task (mediating variable) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A behavioral task assessing attention bias toward positive and negative stimuli. Negative and positive attention bias indices will serve as dependent variables.
Change in baseline Scrambled Sentences Task (mediating variable) scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  A behavioral task assessing interpretation bias toward positive and negative stimuli. Negative and positive interpretation bias indices will serve as dependent variables
CERQ - Acceptance, Rumination, and Reappraisal (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring use of only three emotion regulation strategies
FoC - Fear of Expressing Compassion for Others (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring how much people fear expressing compassion towards others
FoC - Fear of Expressing Kindness and Compassion Towards Oneself (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring how much people fear expressing compassion towards self
S-SCS - Self-kindness (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring levels of kindness shown towards self
S-SCS - Common Humanity (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring feelings of shared humanity
Five Facet Mindfulness Questionnaire (FFMQ; explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring mindfulness on 5 different sub scales. 1 item with the highest factor loading on each of the 5 subscales.
Stress Assessment Questions | Assessed weekly during the course of 10 weeks of intervention only in intervention groups in the context of a stressor
  A scale assessing the occurrence and nature of a stressor
Inclusion of Other in the Self Scale | Assessed weekly during the course of 10 weeks of intervention only in intervention groups in the context of a stressor
  A scale assessing sense of belonging and social connectedness
Frequency and quality of social interaction, and empathic listening | Assessed weekly during the course of 10 weeks of intervention only in intervention groups in the context of a stressor
  A scale assessing quality of social interactions and listening
Penn State Worry Questionnaire (PSWQ)-3 (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring levels of worry
IRI - Personal Distress (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring levels of personal distress felt when showing empathic concern
MAIA - Self-Regulation and Body Listening (explanatory mechanisms) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring levels of interoceptive awareness
Cognitive Control and Flexibility Questionnaire (CCFQ) - Cognitive Control over Emotions (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring cognitive control exhibited over emotional material
Acceptance and Action Questionnaire (AAQ)-II (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring psychological flexibility
DERS (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  1 item each from the following subscales: Nonacceptance of emotional responses, Difficulty engaging in Goal-directed behavior, Lack of emotional awareness, Limited access to emotion regulation strategies, Lack of emotional clarity.
Brief-COPE (explanatory mechanism) | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring the frequency of 2 coping strategies used - emotional support and instrumental support
PSS-4 | Assessed weekly during the course of 10 weeks of intervention only in intervention groups
  A scale measuring perceived stress
Affect Grid (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the intervention groups, prior to and after the daily exercise
  Assessment of emotional state (valence) and arousal
Cube of Thoughts (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the intervention groups, prior to and after the daily exercise
  A scale measuring the temporality and valence of thoughts
Interoception (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the intervention groups, prior to and after the daily exercise
  Assessment of how much bodily sensations are felt
Engagement (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the intervention groups, only once after the daily exercise
  Assessment of how engaged participants felt in the exercise
Social connectedness - Inclusion of Other in Self Scale (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the AD intervention group, prior to and after the daily exercise
  Assessment of how connected participant felt to the dyad partner
Personal Detail Shared (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the AD intervention group, only after the daily exercise
  Assessment of the level of personal details shared by the participant during exercise
Loneliness (explanatory mechanism) | Assessed for 10 weeks during intervention period, 3 times a week, only in the intervention groups, prior to and after the daily exercise
  Assessment of the level of loneliness by the participant before and after exercise
Change from baseline Inflammation Marker levels at 10 weeks | Assessed at pre-test (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Assessment of C-reactive protein (CRP) levels through saliva sample
Change from baseline Polyepigenetic risk scores at 10 weeks | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints only in intervention groups
  Assessment of epigenetic markers through saliva
Belonging to COVID-19 biological risk group | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Belonging to COVID-19 professional risk group | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Positive test result for COVID-19 | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Presence of COVID-19 symptoms | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Hospitalization due to COVID-19 | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Duration of hospitalization due to COVID-19 (in weeks) | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Number of weeks
History of or current presence of long-covid symptoms | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No
Status of COVID-19 vaccination | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  received none, first or both doses
Perception of benefits of COVID-19 vaccination | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  in case of one or two doses received willingness to receive COVID-19 vaccination (in case of no dose received), and impact of COVID-19 related restrictions and limitations
Willing to receive COVID-19 vaccination | Assessed at pre-intervention (Baseline) and then after 10-week intervention period at post-intervention timepoints
  Yes or No. Only in case of no dose received

OTHER OUTCOMES:
TAS-20 (pre-screening) | Assessed prior to the intervention, only once, to pre-screen out from the study individuals who have high levels of alexithymia
  A scale assessing alexithymia
PHQ-9 (pre-screening) | Assessed prior to the intervention, only once, to pre-screen out from the study individuals who have clinical levels of depressive symptoms
  A scale assessing depression
GAD-7 (pre-screening) | Assessed prior to the intervention, only once, to pre-screen out from the study individuals who have clinical levels of anxious symptoms
  A scale assessing generalized anxiety
Standardized Assessment of Personality - Abbreviated Scale (pre-screening) | Assessed prior to the intervention, only once, to evaluate presence of personality disorders
  A self-report scale used to screen personality disorders
Composite International Diagnostic Screener CID-S (pre-screening) | Assessed prior to the intervention, only once, to pre-screen out from the study individuals endorsing clinical levels of psychological disorders
  A self-report scale used to screen mental health

CONTACTS AND LOCATIONS:
Overall Officials: Tania Singer, PhD, Principal Investigator — Social Neuroscience Lab, Max Planck Society
Locations (1):
- Social Neuroscience Lab, Berlin, Germany

REFERENCES:
- [Derived] Silveira S, Godara M, Singer T. Boosting Empathy and Compassion Through Mindfulness-Based and Socioemotional Dyadic Practice: Randomized Controlled Trial With App-Delivered Trainings. J Med Internet Res. 2023 Jul 26;25:e45027. doi: 10.2196/45027. PMID 37494106
- [Derived] Godara M, Silveira S, Matthaus H, Heim C, Voelkle M, Hecht M, Binder EB, Singer T. Investigating differential effects of socio-emotional and mindfulness-based online interventions on mental health, resilience and social capacities during the COVID-19 pandemic: The study protocol. PLoS One. 2021 Nov 4;16(11):e0256323. doi: 10.1371/journal.pone.0256323. eCollection 2021. PMID 34735441